CLINICAL TRIAL: NCT02966847
Title: Assessment of Cone-beam Computed Tomography (CBCT) Assistance to Video-assisted Thoracoscopic Surgery
Acronym: CAVIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 35RC16_9838; 2016-A01353-48 (Other: Id-RCB)
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Thoracoscopy
Keywords: Video assisted thoracoscopy; Cone beam computed tomography
MeSH Terms: interventions — Anesthesia; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBCT Acquisition (Experimental): The anesthesia and surgery will take place in the usual way. The intervention consists in the CBCT acquisition after the initiation of single-lung ventilation, after the introduction of trocars.
  Interventions: Procedure: CBCT acquisition; Procedure: Anesthesia and surgery

INTERVENTIONS:
Procedure: CBCT acquisition — Acquisitions are performed with the DynaCT function of a C-arm Artis Zeego System® device
  Other Names: Artis Zeego System®
Procedure: Anesthesia and surgery — The anesthesia and surgery will take place according clinical routine practice

SUMMARY:
In the coming years, an increase in lung nodule resection is expected, particularly in Video-assisted thoracoscopic surgery (VATS). In some situations, it is necessary to use a device for locating these nodules. Meanwhile, the Cone Beam Computed Tomography (CBCT) is a tool whose use is constantly spreading.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the feasibility of using intraoperative CBCT to develop a new procedure for intraoperative localization of pulmonary nodules in video-assisted thoracoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18;
* patient with unique or multiple pulmonary lesions of a size ranging from 5 to 20 mm;
* Complete preoperative assessment;
* Patient receiving information about the protocol who did not indicate his/her opposition to participate;
* Patient covered by a social insurance system

Exclusion Criteria:

* Reoperation (history of ipsilateral thoracic surgery);
* Inability to achieve or obtain a single-lung ventilation during surgery;
* Adult subject to legal protection (trusteeship, guardianship);
* Person deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Assessment of CBCT | the day following the acquisition
  Ability to identify the lesion on CBCT images of unventilated lung. CBCT images are interpreted by 2 senior surgeons.

SECONDARY OUTCOMES:
Feasibility of CBCT | At the end of the surgery
  Number of patient excluded because of an inability to achieve CBCT acquisition, whatever the reason.
Assessment of global image quality | the day following the acquisition
  Assessment of image quality is based on an "open label" interpretation of CBCT images by two senior surgeons who score images from 0 (uninterpretable) to 10 (same quality as CT images)
Assessment of image quality of lesions | the day following the acquisition
  Assessment of image quality depending on the type of lesion and their location. Interpretation of CBCT images are performed by two senior surgeons who score images from 0 (uninterpretable) to 10 (same quality as CT images)

CONTACTS AND LOCATIONS:
Overall Officials: Simon ROUZE, MD, Principal Investigator — CHU Rennes
Locations (1):
- Centre Hospitalier Universitaire de RENNES, Rennes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alvarez P, Rouze S, Miga MI, Payan Y, Dillenseger JL, Chabanas M. A hybrid, image-based and biomechanics-based registration approach to markerless intraoperative nodule localization during video-assisted thoracoscopic surgery. Med Image Anal. 2021 Apr;69:101983. doi: 10.1016/j.media.2021.101983. Epub 2021 Jan 30. PMID 33588119